CLINICAL TRIAL: NCT01197417
Title: Intravenous Magnesium for Sickle Cell Vasoocclusive Crisis
Acronym: MAGiC
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: Pediatric Emergency Care Applied Research Network (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PECARN 025
Record Dates: First submitted 2010-08-31; First posted 2010-09-09 (Estimated); Results first posted 2015-09-07 (Estimated); Last update posted 2016-01-27 (Estimated); Status verified 2015-12

CONDITIONS: Sickle Cell Disease
Keywords: Sickle Cell Disease; Magnesium Sulfate; Pediatric
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Magnesium group (Experimental): Intravenous Magnesium Sulfate
  Interventions: Drug: Intravenous Magnesium Sulfate
- Placebo group (Placebo Comparator): Normal Saline placebo
  Interventions: Drug: Normal Saline Placebo

INTERVENTIONS:
Drug: Intravenous Magnesium Sulfate — 40 mg/kg (max 2.4 grams), infused at a concentration of 40 mg/ml (1 ml/kg, max 60 ml), every 8 hours for a total of 6 doses
  Arms: Magnesium group
Drug: Normal Saline Placebo — (1 ml/kg, max 60 ml), administered every 8 hours for a total of 6 doses
  Arms: Placebo group

SUMMARY:
The purpose of this study is to determine the safety and efficacy of intravenous magnesium in shortening the duration of a pain crisis and to determine the health-related quality of life and short term outcomes of children treated with intravenous magnesium during an acute pain crisis.

DETAILED DESCRIPTION:
It is well known that children with sickle cell disease are at risk for acute pain crises. The usual treatment for these pain crises, intravenous fluids and pain medicines such as morphine, has changed little over the past three decades. In a pilot study, the addition of intravenous magnesium to standard therapy decreased length of stay; however, this study was not randomized, not blinded, not placebo-controlled, and not adequately powered to assess safety.

We will conduct a multi-center, randomized, double-blind, placebo controlled trial of about 208 children, ages 4-21 years. Patients will be randomized to receive intravenous magnesium sulfate or placebo every 8 hours for a total of 6 doses, or until discharge. Patients will return for a routine clinic visit up to 3 months after discharge for a baseline assessment. Patients will also complete health-related quality of life measures at 4 timepoints throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* age 4-21 years, inclusive
* Sickle cell anemia (Hb SS) or Sickle beta zero thalassemia disease (Hb Sβ°)
* failed intravenous opioid pain management in the emergency department prior to the decision to admit the patient
* admitted to the inpatient unit for sickle cell pain crisis

Exclusion Criteria:

* patient received more than 12 hours of intravenous pain medication prior to enrollment
* previous enrollment in this study (only one admission per child is eligible)
* history of allergy/intolerance to both intravenous morphine and hydromorphone
* known other cause for pain (avascular necrosis, gall bladder disease, priapism, etc.)
* patient with greater than 10 admissions for pain crisis in the past year
* patient maintained on daily opioids or chronic transfusions for chronic sickle cell pain
* transfusion within the previous two months
* known kidney or liver failure (elevation of liver function tests does not warrant exclusion)
* known pulmonary hypertension
* pregnancy
* diagnosis of bacterial infection, fever ≥39.5°C, acute chest syndrome, hemodynamic instability or sepsis
* current oral magnesium supplementation or current enrollment in another therapeutic study protocol
* previously diagnosed clinical stroke
* current or planned use of neuromuscular blocker, nifedipine, ritodrine, or terbutaline
* allergy to magnesium sulfate
* discharge from an inpatient unit within 72 hours of arrival in the emergency department for the current pain crisis

Ages: 4 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 208 (Actual)
Dates: Start 2010-12; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Brousseau, MD, MS, Principal Investigator — Medical College of Wisconsin
Locations (8):
- United States (8):
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Children's Hospital of Michigan, Detroit, Michigan
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital of Philadelphia Research Institute, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Baylor College of Medicine, Houston, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Result] Brousseau DC, Scott JP, Badaki-Makun O, Darbari DS, Chumpitazi CE, Airewele GE, Ellison AM, Smith-Whitley K, Mahajan P, Sarnaik SA, Casper TC, Cook LJ, Dean JM, Leonard J, Hulbert ML, Powell EC, Liem RI, Hickey R, Krishnamurti L, Hillery CA, Nimmer M, Panepinto JA; Pediatric Emergency Care Applied Research Network (PECARN). A multicenter randomized controlled trial of intravenous magnesium for sickle cell pain crisis in children. Blood. 2015 Oct 1;126(14):1651-7. doi: 10.1182/blood-2015-05-647107. Epub 2015 Jul 31. PMID 26232172
- [Derived] Panepinto JA, Paul Scott J, Badaki-Makun O, Darbari DS, Chumpitazi CE, Airewele GE, Ellison AM, Smith-Whitley K, Mahajan P, Sarnaik SA, Charles Casper T, Cook LJ, Leonard J, Hulbert ML, Powell EC, Liem RI, Hickey R, Krishnamurti L, Hillery CA, Brousseau DC; Pediatric Emergency Care Applied Research Network (PECARN). Determining the longitudinal validity and meaningful differences in HRQL of the PedsQL Sickle Cell Disease Module. Health Qual Life Outcomes. 2017 Jun 12;15(1):124. doi: 10.1186/s12955-017-0700-2. PMID 28606098
- [Derived] Badaki-Makun O, Scott JP, Panepinto JA, Casper TC, Hillery CA, Dean JM, Brousseau DC; Pediatric Emergency Care Applied Research Network (PECARN) Magnesium in Sickle Cell Crisis (MAGiC) Study Group. Intravenous magnesium for pediatric sickle cell vaso-occlusive crisis: methodological issues of a randomized controlled trial. Pediatr Blood Cancer. 2014 Jun;61(6):1049-54. doi: 10.1002/pbc.24925. Epub 2014 Jan 17. PMID 24443249

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Magnesium Group | Placebo Group
Started | 104 | 104
Received Study Drug | 101 | 103
Completed | 96 | 86
Not Completed | 8 | 18
Not completed — Physician Decision | 3 | 2
Not completed — Withdrawal by Subject | 2 | 4
Not completed — Site miscommunication | 0 | 1
Not completed — Subject transferred to intensive care | 0 | 1
Not completed — Not consented in time to receive drug | 0 | 1
Not completed — Hypotension | 1 | 2
Not completed — Found to be ineligible | 2 | 5
Not completed — No 25-hour magnesium level | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Magnesium Group | Placebo Group | Total
Number analyzed (Participants) | 104 | 104 | 208
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 93 | 88 | 181
  Between 18 and 65 years | 11 | 16 | 27
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.4 (4.5) | 13.8 (4.8) | 13.6 (4.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 57 | 108
  Male | 53 | 47 | 100
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 5 | 8
  Not Hispanic or Latino | 96 | 94 | 190
  Unknown or Not Reported | 5 | 5 | 10
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Pacific Islander | 0 | 0 | 0
  Black or African American | 99 | 94 | 193
  White | 0 | 0 | 0
  More than one race | 2 | 3 | 5
  Unknown or not reported | 3 | 4 | 7
  Other | 0 | 3 | 3
Region of Enrollment [Number; unit: participants]
  United States | 104 | 104 | 208

OUTCOME MEASURES:

1. Primary Outcome: Hospital Length of Stay (Hours)
Time Frame: From the time of the start of first study med infusion until hospital discharge or 12 hours after the last IV opioid, whichever occurs first, up to 10 days post enrollment
Population: All participants who received at least one dose of study drug and who did not withdraw from data collection prior to outcome
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Magnesium Group | Placebo Group
Number analyzed (Participants) | 100 | 102
hours | 56 [27 to 109] | 47 [24 to 99]
Statistical Analysis 1: Comparison: Magnesium Group vs Placebo Group; Null hypothesis of equal distributions of primary length of stay between treatment arms within all randomization strata; Test type: Superiority or Other; p = 0.24, Van Elteren test; Randomization strata were defined by enrollment site, age group and hydroxyurea use within the last three months prior to enrollment

2. Secondary Outcome: Number of Morphine Equivalents Per Kilogram of Body Weight Used During Hospitalization
Time Frame: Total morphine equivalents used during the hospitalization will be recorded on the day of discharge, up to 10 days post enrollment
Population: All participants who received at least one dose of study drug and who did not withdraw from data collection prior to either hospital discharge or 12 hours after last intravenous opioid.
Measure: Median (Inter-Quartile Range); unit: mg Morphine/kg
Arm/Group | Magnesium Group | Placebo Group
Number analyzed (Participants) | 100 | 102
mg Morphine/kg | 1.46 [0.55 to 3.32] | 1.28 [0.40 to 3.29]
Statistical Analysis 1: Comparison: Magnesium Group vs Placebo Group; Test type: Superiority or Other; p = 0.12, Van Elteren test; [statistical method as in outcome 1, analysis 1]

3. Secondary Outcome: Hypotension Associated With Infusion
Description: For each study drug infusion, systolic blood pressure (SBP) was measured just prior to the start of the infusion and again every 10 minutes until 30 minutes until the end of the infusion. Hypotension was defined as a greater than 20% reduction in SBP relative to corresponding baseline measurement for any study drug infusion.
Time Frame: Blood pressure will be monitored every 8 hours, concurrent with each infusion, and for 20-30 minutes after infusion completion, until discharge, up to 2 days post enrollment
Population: All participants who received at least one dose of study drug
Measure: Number; unit: Participant
Arm/Group | Magnesium Group | Placebo Group
Number analyzed (Participants) | 101 | 103
Participant | 4 | 1
Statistical Analysis 1: Comparison: Magnesium Group vs Placebo Group; Test type: Superiority or Other; p = 0.39, Mantel Haenszel; [statistical method as in outcome 1, analysis 1]

4. Secondary Outcome: Warm Sensation Associated With Study Drug Infusion
Description: Patient spontaneously reported feelings of warmth during any study drug infusion.
Time Frame: Patient-reported warm sensation upon infusion will be monitored every 8 hours, concurrent with each infusion, and for 20-30 minutes after infusion completion, until discharge, up to 2 days post enrollment
Population: All participants who received at least one dose of study drug.
Measure: Number; unit: Participant
Arm/Group | Magnesium Group | Placebo Group
Number analyzed (Participants) | 101 | 103
Participant | 26 | 2
Statistical Analysis 1: Comparison: Magnesium Group vs Placebo Group; Test type: Superiority or Other; p < 0.01, Mantel Haenszel; [statistical method as in outcome 1, analysis 1]

5. Secondary Outcome: Rehospitalization
Time Frame: Rehospitalization will be measured at 7 days post discharge and at the follow-up visit (on average, 30 days post discharge)
Population: All participants who received at least one dose of study drug who had known rehospitalization status within 7 days
Measure: Number; unit: Participant
Arm/Group | Magnesium Group | Placebo Group
Number analyzed (Participants) | 100 | 102
Participant | 12 | 7
Statistical Analysis 1: Comparison: Magnesium Group vs Placebo Group; Test type: Superiority or Other; p = 0.11, Mantel Haenszel; [statistical method as in outcome 1, analysis 1]

6. Secondary Outcome: Development of Acute Chest Syndrome (ACS)
Time Frame: Patients will be monitored daily, on average, during their length of stay until discharge, up to 10 days post enrollment
Measure: Number; unit: Paricipants
Arm/Group | Magnesium Group | Placebo Group
Number analyzed (Participants) | 101 | 103
Paricipants | 16 | 14
Statistical Analysis 1: Comparison: Magnesium Group vs Placebo Group; Test type: Superiority or Other; p = 0.78, Van Elteren test; [statistical method as in outcome 1, analysis 1]

7. Secondary Outcome: Hospital Length of Stay
Time Frame: Start of first study drug infusion to actual hospital discharge
Measure: Median (Inter-Quartile Range); unit: Hours
Arm/Group | Magnesium Group | Placebo Group
Number analyzed (Participants) | 100 | 102
Hours | 74.5 [39.5 to 123.5] | 60.5 [37 to 122]
Statistical Analysis 1: Comparison: Magnesium Group vs Placebo Group; Test type: Superiority or Other; p = 0.46, Van Elteren test; [statistical method as in outcome 1, analysis 1]

ADVERSE EVENTS:
Description: Participant Flow and Baseline characteristics are reported for all randomized patients; however, adverse events only include the 204 (98%) who received study drug.
Groups:
- Magnesium Group: Intravenous Magnesium Sulfate Intravenous Magnesium Sulfate: 40 mg/kg (max 2.4 grams), infused at a concentration of 40 mg/ml (1 ml/kg, max 60 ml), every 8 hours for a total of 6 doses
- Placebo Group: Normal Saline placebo Normal Saline Placebo: (1 ml/kg, max 60 ml), administered every 8 hours for a total of 6 doses
Arm/Group | Magnesium Group | Placebo Group
Serious Adverse Events (participants affected / at risk) | 13/101 | 12/103
Other Adverse Events (participants affected / at risk) | 66/101 | 62/103
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Magnesium Group (N=101) | Placebo Group (N=103)
Acute chest syndrome (Blood and lymphatic system disorders) | 10 (10) | 7 (7)
Gallstones (Hepatobiliary disorders) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Decreased hemoglobin (Investigations) | 0 (0) | 4 (4)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Magnesium Group (N=101) | Placebo Group (N=103)
Acute chest syndrome (Blood and lymphatic system disorders) | 6 (6) | 7 (7)
Anemia (Blood and lymphatic system disorders) | 7 (7) | 7 (7)
Constipation (Gastrointestinal disorders) | 8 (8) | 11 (11)
Emesis (Gastrointestinal disorders) | 10 (10) | 9 (9)
Nausea (Gastrointestinal disorders) | 16 (16) | 19 (20)
Vomiting (Gastrointestinal disorders) | 5 (5) | 11 (11)
Fever (General disorders) | 27 (31) | 26 (26)
Warmth (General disorders) | 8 (10) | 0 (0)
Oxygen saturation decreased (Investigations) | 8 (8) | 12 (12)
Dizziness (Nervous system disorders) | 6 (7) | 4 (4)
Headache (Nervous system disorders) | 12 (13) | 9 (11)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 6 (6)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 2 (2)
Itching (Skin and subcutaneous tissue disorders) | 12 (12) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No